CLINICAL TRIAL: NCT04930068
Title: Ultrasonic Cavitation on Abdominal Obesity in Adolescent Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Ghada ebrahim El Refaye - Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Cairo University, Egypt (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo Un112
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Ultrasonic
Keywords: Ultrasonic; aerobic exercise; Diet
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Group (A) consisted of 25 females who treated by ultrasonic cavitation, group (B) consisted of 25 females who performed aerobic exercise.
Who Masked: Outcomes Assessor
Masking Description: closed enveloped
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra-sound (Experimental): ultrasonic cavitation applied on abdominal region for 30 minutes, 2 times per week for 6 weeks.
  Interventions: Other: low caloric diet
- aerobic exercise (Experimental): aerobic exercises through treadmill (60-70% of VO2 max.) for 30 minutes, 2 times per week for 6 weeks
  Interventions: Other: low caloric diet

INTERVENTIONS:
Other: low caloric diet — A low-calorie diet is a structured eating plan that restricts daily caloric intake, commonly for weight loss. Following a low-calorie diet typically means consuming around 1,200 to 1,500 calories per day, which creates a calorie deficit that can lead to weight loss. A low-calorie diet can be effective, but it requires a lot of discipline to work and be safe.

SUMMARY:
The purpose of this study was to determine the effect of ultrasonic cavitation on abdominal obesity in females. Fifty volunteer females with abdominal obesity participated in the study.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effectiveness of ultrasonic cavitation on abdominal obesity in adolescent females. Fifty volunteer females with abdominal obesity participated in the study.

Group (A) consisted of 25 females who treated by ultrasonic cavitation on abdominal region for 30 minutes and aerobic exercises for 30 minutes, 2 times per week for 6 weeks ; group (B) consisted of 25 females who performed aerobic exercise and low caloric diet.

ELIGIBILITY:
Inclusion Criteria:

* Their ages were range from 17 to 21 years old.
* Their body mass index less than 35kg/m2.

Exclusion Criteria:

* Females with BMI exceed 35kg/m2.
* Females have psychological disorders.
* cardiac diseases.
* hypertension

Ages: 17 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Bioelectrical impedance analysis | 6 weeks
  was used to estimate body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Most body water is stored in muscle in both groups A and B

SECONDARY OUTCOMES:
skin fold caliper | 6 weeks
  was used to measure the waist circumference and amount of subcutaneous fat when the fold for all females in both groups (A&B)

CONTACTS AND LOCATIONS:
Overall Officials: Ghada E Elrefaye, professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy- Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No